CLINICAL TRIAL: NCT01772342
Title: Effects of a Novel Purifying Device (PureNight) on Sleep Quality in Chronic Obstructive Pulmonary Disease
Brief Title: Effects of an Air Purifying Device (PureNight) on Sleep Quality in Obstructive Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miriam D Cohen, Nurse Practitioner, VA New York Harbor Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01056
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Sleep Fragmentation; Quality of Life; Air Filters
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Deprivation | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nocturnal Air Purification (Experimental): * Hepa Filtration with PureNight
  * SHAM with PureNight
  Interventions: Other: HEPA filtration; Other: SHAM

INTERVENTIONS:
Other: HEPA filtration — Night time air purification with the PureNight air purification system with the HEPA filter in place
Other: SHAM — Night time air purification with the PureNight air purification system with the HEPA filter removed

SUMMARY:
Many individuals with chronic lung disease have night time symptoms that disrupt their sleep. The purpose of this study is to determine the effects of an air purifying device (PureNight, Halo Innovations, Minneapolis, MN) on sleep disruptions measured by a "sleep watch" (actigraph) and individual perception of sleep quality.

DETAILED DESCRIPTION:
Objective There are many detrimental effects of obstructive airway disease. One of the hallmark effects is poor sleep quality. Due to the association of air pollutants with worsening respiratory symptoms, a logical intervention to improve sleep quality may be air filtration. A novel air filtration system, the PureNight SystemTM, which delivers pre-filtered air around the head of a sleeping person, may offer a solution to decrease exposure to noxious triggers during time spent sleeping and improve sleep quality.

One method to measure sleep quality is to use 24-hour actigraphy. The actigraph is a small, wrist-worn device that contains a pizo-electric bender element, or accelerometer, that measures wrist movement. Algorithms interpret the movement on an epoch-by-epoch basis and identify sleep/wake states and circadian rhythms from activity counts.

Study Design We propose to study the effect of the Pure Night TM air filtration system on a cohort of patients with chronic obstructive airway disease with self-reported poor sleep quality due to nocturnal respiratory symptoms. We hypothesized that patients using the Pure Night TM system would have fewer nocturnal awakenings and a consolidation of sleep time measured by actigraphy and better sleep quality measured by quality of sleep questionnaires than when not using the device. In a cross-over randomized clinical trial, baseline measurements were compared to treatment with the PureNight TM device and with "sham" filtration. Sleep variables including data on circadian rhythms were compared using a within-subject design between test conditions.

Methodology Each subject underwent baseline actigraphy over 7 days followed by two seven day treatment arms with a 7-day wash-out period between treatment arms. Subject slept with the PureNight during each arm of the study. The systems used in each arm of the study were identical except one arm had a sham filter replacing the HEPA filter of the PureNight TM system in random order. Participants completed the Pittsburgh Sleep Quality Index at the start of the study and at the end of each treatment phase. Objective estimates of sleep were calculated from the actigraphy recordings using the device's proprietary software.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD, chronic airway obstruction, chronic bronchitis or emphysema or > 15 pack year history of tobacco use
* Secondary diagnosis of extrinsic asthma or allergic rhinitis or > 200 ml FEV1 response to bronchodilators documented on pulmonary function testing
* Positive score on sleep quality questionnaire

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Impairment of cognition or communication
* History of drug or alcohol treatment within the past 6 months
* Recent acute medical event that would suggest a contraindication to participate at the scheduled time
* Treatment with antibiotics or steroids for COPD exacerbation within past 6 weeks
* Baseline of three or more episodes of nocturia per night
* On home oxygen or non-invasive positive pressure breathing
* Diagnosis of obstructive sleep apnea or body mass index > 35
* Primary sleep disorder, such as insomnia

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Fragmentation Index from baseline | Measurements are averaged during the first week of the study (baseline) and then during week 2 and week 4 when subjects slept with the air purifier with either HEPA or SHAM filtration
  Data is obtained from a wrist-worn motion sensor that detects body movement. From these data, the number of disruptions during sleep can be calculated.

SECONDARY OUTCOMES:
Change in Sleep-related quality of life from baseline | Measurements are taken at the start of the study (baseline) and then at the end of week 2 and week 4 when subjects slept with the air purifier with either HEPA or SHAM filtration
  Total score of Pittsburgh Sleep Quality Index, which is a health-related quality of sleep questionnaire that measures perception of sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Miriam D Cohen, Principal Investigator — VA, NYHH